CLINICAL TRIAL: NCT06893406
Title: Cervical Myelopathy in Hip Fracture Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Jamie Bradbury, Associate Professor of Clinical Neurological Surgery, Indiana University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: 24990
Record Dates: First submitted 2025-03-18; First posted 2025-03-25 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Cervical Myelopathy; Hip Fractures
Keywords: Hip fracture; Cervical myelopathy
MeSH Terms: conditions — Hip Fractures | interventions — Health Records, Personal; Restraint, Physical

STUDY DESIGN:
Intervention Model Description: All hip fracture patients that provide consent for participation will undergo a history and physical examination to specifically evaluate for potential cervical myelopathy. If the history and physical exam detect signs or symptoms of cervical myelopathy, a cervical MRI will be scheduled to confirm the diagnosis.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation for Cervical Myelopathy (Experimental): Hip fracture patients who agree to participate will undergo a history and physical exam to specifically evaluate for clinical signs or symptoms of cervical myelopathy. If the history and physical exam is positive for such symptoms, a cervical MRI will be scheduled as part of standard care to further evaluate for this diagnosis. If the history and physical exam is negative for such symptoms, further clinical evaluation for this condition will not occur.
  Interventions: Diagnostic Test: Cervical MRI; Other: History & Physical Exam

INTERVENTIONS:
Diagnostic Test: Cervical MRI — Participants whose history and physical exam indicate signs or symptoms of cervical myelopathy will be scheduled for a cervical MRI.
Other: History & Physical Exam — A history and physical exam to evaluate for specific signs and symptoms of cervical myelopathy will be performed.

SUMMARY:
Recent evidence has demonstrated a high rate of undiagnosed cervical myelopathy in patients presenting with hip fractures from a ground level fall. Identification and treatment of cervical myelopathy can help prevent falls and future fragility fractures. The purpose of this study is to screen ground level fall hip fracture patients for cervical myelopathy using a history, physical exam, and then offer an MRI if indicated.

DETAILED DESCRIPTION:
Cervical myelopathy is compression of the cervical spinal cord which causes many things, but a common and prominent symptom is poor coordination/balance. This has been shown in multiple high quality studies to increase a patient's risk of falls as well as fragility fractures (such as hip fractures). Often, patients with hip fractures present with multiple falls of unknown origin. Work up from an orthopedic perspective is rare, but our medicine colleagues spend a substantial amount of resources to identify a cause (carotid ultrasound, head CT, EKG, echo, labs, etc.). This is because hip fractures in the elderly come with a 10-30% risk of death at one year. Preventing a fall that causes a hip fracture is very important, and we, as orthopedists, are well positioned to aid in that endeavor. 8 years ago a study was published in a prominent orthopedic journal looking at cervical myelopathy in hip fracture patients. With 28 hip fracture patients, they found an 18% rate of cervical myelopathy. This was diagnosed on history and physical exam. MRIs were offered but not obtained. To date, this is the only study on this subject. This study will be similar but will go a step further and obtain a cervical spine MRI to complete the diagnosis of cervical myelopathy for these patients. This can help get them on the pathway for treatment and future fall prevention.

How it will work:

Once a patient sustains a hip fracture and is admitted to either Methodist hospital, IU North hospital, or Eskenazi hospital, study team will screen the patient for inclusion and exclusion criteria via chart review. If criteria are met, the patient will be seen in the hospital by study team and the patient will be consented for the study. The study team will do a physical exam and take a history from the patient for research purposes, looking for signs/symptoms of cervical myelopathy. If it is determined the patient likely has cervical myelopathy, as standard of care, the patient will be offered an MRI and possibly be referred to a surgeon.

ELIGIBILITY:
Inclusion Criteria:

* Patient admitted to Eskenazi, Methodist, or IU North hospital for a hip fracture (femoral neck, intertrochanteric, subtrochanteric, or pertrochanteric fracture) that was caused by a ground level fall.

Exclusion Criteria:

* Neurologic or cognitive disorder explaining the fall (dementia, Parkinson's disease, delirium, etc.)
* Syncopal fall or fall caused by stroke or a heart condition

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-03-20 (Estimated)

PRIMARY OUTCOMES:
Detection of cervical myelopathy on history and physical exam | Once, at time of enrollment
  The number of hip fracture participants whose history and physical exam positively demonstrate signs or symptoms of cervical myelopathy will be compared to the number of hip fracture participants whose history and physical exam do not demonstrate signs or symptoms of cervical myelopathy.
Diagnosis of cervical myelopathy on cervical MRI | Once, prior to hospital discharge
  Hip fracture participants whose history and physical exam positively demonstrate signs or symptoms of cervical myelopathy will be referred for a cervical MRI, to occur prior to hospital discharge. The number of participants whose cervical MRI confirms this diagnosis will be compared to the number of participants for whom cervical MRI does not confirm this diagnosis.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Indiana University North Hospital, Fishers, Indiana
  - Eskenazi Hospital, Indianapolis, Indiana
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Radcliff KE, Curry EP, Trimba R, Walker JB, Purtill JJ, Austin MS, Parvizi J, Vaccaro AR, Hilibrand AS, Albert TJ. High Incidence of Undiagnosed Cervical Myelopathy in Patients With Hip Fracture Compared With Controls. J Orthop Trauma. 2016 Apr;30(4):189-93. doi: 10.1097/BOT.0000000000000485. PMID 26562581